CLINICAL TRIAL: NCT02485223
Title: Single Test to ARrive at MS Diagnosis. A Prospective, Longitudinal, Investigator Blinded, Pilot Study Assessing the Accuracy of a Single 3 Tesla MRI Scan in Predicting Multiple Sclerosis in Cases of Diagnostic Uncertainty
Brief Title: Single Test to ARrive at MS Diagnosis. Using a Single MRI Brain Scan to Help Diagnose Multiple Sclerosis
Acronym: STAR-MS
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 15022 [Sponsor reference]; 15/NW/0286 (Other: NRES Committee North West - Greater Manchester East)
Record Dates: First submitted 2015-04-23; First posted 2015-06-30 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; MS; Diagnostic test; Central veins; MRI
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a pilot study (a small scale study testing procedures so that the investigators can apply this to a larger scale study). This study will test the accuracy of a new brain scan (Magnetic Resonance Imaging) technique in predicting the diagnosis of multiple sclerosis (MS) in patients where there is uncertainty about the diagnosis. For patients where there is a suspicion (but not definite) diagnosis of MS, an additional MRI brain scan will be offered. There will be no other research tests and the patient is followed up to see what the eventual diagnosis is. The investigators will then review the original brain scan to see if this predicted the diagnosis of MS or not.

DETAILED DESCRIPTION:
There is no single, simple test to differentiate MS from conditions that mimic it. Apart from the patient's symptoms, doctors use Magnetic Resonance Imaging (MRI) of the brain to see if there are abnormalities which are consistent with MS. In patients without typical symptoms or a typical MRI appearance, a firm diagnosis cannot be made as other neurological illnesses can mimic symptoms of MS and the MRI scans can look very similar. Further tests are often required such as lumbar punctures, resulting in delays, discomfort for the patient and additional healthcare costs. With time the diagnosis can become clearer as patients may develop other symptoms of MS but this may take months or years.

The most common errors are from misinterpretation of the brain abnormalities or 'lesions' seen on the MRI scan. Subsequently if a patient is misdiagnosed with MS they may receive treatment they do not need. Furthermore a delay in a firm diagnosis delays treatment for another condition. With the rapid increase of new medications in the last few years, accurate and rapid diagnosis is paramount.

Pathologically (when looking at lesions using a microscope) MS lesions usually have a vein running through the centre, whereas in lesions arising from other conditions, the investigators hypothesize that no central vein is seen. The investigators can therefore distinguish between patients with MS and patients without it.

The researchers therefore want to test the value of a clinical 3-Tesla MRI brain scan in accurately distinguishing between MS and other conditions, with MRI sequences that have been refined over the last few years.

Patients will only have one research MRI brain scan and then be followed up by their neurologist, who will confirm the final diagnosis. The investigators shall then look back at the original scans to see if those with MS had veins within their lesions and if those without MS had lesions without veins

ELIGIBILITY:
Inclusion Criteria:

* Able to tolerate an MRI brain scan
* No contraindications to MRI
* Radiological suspicion of MS, but clinically atypical or Clinical suspicion of MS, but radiologically atypical
* Radiological or clinical suspicion of any of the following with a routine MRI brain scan showing white matter lesions; Autoimmune/Inflammatory; Antiphospholipid syndrome, Neurosarcoidosis, Neuro-Behcet's disease, Neuromyelitis Optica, Systemic lupus erythematosus, Primary CNS vasculitis, Secondary CNS vasculitis, Sjogren's syndrome, Susac syndrome. Ischaemic; Hypertensive ischaemic disease (small vessel disease), embolic disease. Infective ; Lyme disease, Cytomegalovirus CNS infection, Toxocariasis, Neurocysticercosis, Whipple's disease, Progressive Multifocal Leukoencephalopathy, Herpes virus (HHV) infection e.g VZV, HIV, Toxoplasmosis, Tuberculosis, Neurosyphilis. Neoplastic; Lymphoma, Glioma, Primary CNS Lymphoma, Cerebral metastases. Other; CADASIL, Histiocytosis, Migraine, Mitochondrial disease, Leukodystrophy.

Exclusion Criteria:

* Unable to tolerate a further MRI scan
* Unsafe to perform an MRI scan
* Pregnancy
* Participants with normal routine clinical scans
* Unable to give written informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators will recruit patients who attend the general neurology and MS clinics at Nottingham University Hospitals (NUH) NHS Trust, UK. The researchers anticipate that the study population will comprise of two groups: the common presentation of young individuals following the first neurological symptoms suggestive of MS, however the neuroradiologist's report of the MRI will not be in agreement with the neurological impression; and a group of patients who present with atypical symptoms for MS but the MRI scan is reported as suggestive of MS.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Difference in the proportion of central veins:lesions in patients with MS and non-MS. | After 1 year of follow up with a confirmed diagnosis.
  To detect this difference with an alpha of 0.05 and power of 0.8, (based on previous data that shows a mean proportion of approx. 60% in MS patients and 6% in ischaemic patients) we will need 12 patients with MS and 12 with non-MS at 1 year of follow up. However given the fact that approx. 40% of patients will have a diagnosis of MS at 1 year, we will need to scan 60 patients in total.

SECONDARY OUTCOMES:
Sensitivity of using a proportion of central veins:lesions in diagnosing MS. | After 1 year of follow up with a confirmed diagnosis
Specificity of using a proportion of central veins:lesions in diagnosing MS. | After 1 year of follow up with a confirmed diagnosis
Positive predictive value of the central vein:lesion MRI test. | After 1 year of follow up with a confirmed diagnosis
Negative predictive value of the central vein:lesion MRI test. | After 1 year of follow up with a confirmed diagnosis
Optimal proportion of central veins:lesions to make a diagnosis of MS. | After 1 year of follow up with a confirmed diagnosis.
  Receiver Operating Characteristic (ROC) curves will be used.
Rate of patient recruitment. | After 1 year
Cohen's kappa inter-rater agreement for the diagnosis of MS using the MRI test. | After 1 year of follow up.
  Can different observers calculate the same proportion of central veins:lesions on each scan.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Nikos Evangelou, MD, Principal Investigator — Clinical Neurology, Division of Clinical Neuroscience, University of Nottingham, UK
Locations (1):
- Clinical Neurology, Division of Clinical Neuroscience, University of Nottingham, UK, Nottingham, Nottinghamshire, United Kingdom

REFERENCES:
- [Background] Tallantyre EC, Brookes MJ, Dixon JE, Morgan PS, Evangelou N, Morris PG. Demonstrating the perivascular distribution of MS lesions in vivo with 7-Tesla MRI. Neurology. 2008 May 27;70(22):2076-8. doi: 10.1212/01.wnl.0000313377.49555.2e. No abstract available. PMID 18505982
- [Background] Tallantyre EC, Dixon JE, Donaldson I, Owens T, Morgan PS, Morris PG, Evangelou N. Ultra-high-field imaging distinguishes MS lesions from asymptomatic white matter lesions. Neurology. 2011 Feb 8;76(6):534-9. doi: 10.1212/WNL.0b013e31820b7630. PMID 21300968
- [Background] Mistry N, Dixon J, Tallantyre E, Tench C, Abdel-Fahim R, Jaspan T, Morgan PS, Morris P, Evangelou N. Central veins in brain lesions visualized with high-field magnetic resonance imaging: a pathologically specific diagnostic biomarker for inflammatory demyelination in the brain. JAMA Neurol. 2013 May;70(5):623-8. doi: 10.1001/jamaneurol.2013.1405. PMID 23529352
- [Background] Sati P, George IC, Shea CD, Gaitan MI, Reich DS. FLAIR*: a combined MR contrast technique for visualizing white matter lesions and parenchymal veins. Radiology. 2012 Dec;265(3):926-32. doi: 10.1148/radiol.12120208. Epub 2012 Oct 16. PMID 23074257